CLINICAL TRIAL: NCT00354653
Title: AN OPEN STUDY OF LAMIVUDINE TREATMENT IN ADULT HBeAg NEGATIVE (Presumed Pre-core Mutant) CHRONIC HEPATITIS B PATIENTS IN IRAN.
Brief Title: A Trial To Study The Effect Of Lamivudine In Adult Patients Who Suffer From Chronic Hepatitis B Alone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NUC 30956
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: CHRONIC HEPATITIS B
Keywords: HBeAg; HBV; CHRONIC HEPATITIS; lamivudine
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis, Chronic | interventions — Lamivudine

INTERVENTIONS:
Drug: LAMIVUDINE

SUMMARY:
The efficacy of lamivudine in Hepatitis Be Antigen (HBeAg) positive Asian patients of chronic hepatitis has been well established.The evidence in HBeAg negative patients is limited. Limited sustained response was observed post-treatment following a one year treatment period. Whether these results can be applied to patients in Iran is uncertain. This study is therefore intended to further assess the efficacy profile after two years of open treatment in the adult Iranian population.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed active liver disease due to Hepatitis B virus.
* Patients must have adequate blood & liver functions.
* Female patients of child-bearing potential must be non pregnant and willing to abstain from intercourse from 2 weeks prior to administration of the first dose of study medication until 28 days after the final dose of study medication or be willing to consistently and correctly use an acceptable method of birth control.
* Patients who have serious concurrent illnesses other than hepatitis B like cancer, severe heart disease, uncontrolled diabetes mellitus or AIDS will not be eligible.

Exclusion Criteria:

* Persons allergic to lamivudine or suffering from hepatitis C, D or E infection or taking alcohol will not be eligible.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2002-02-09 (Actual); Primary Completion 2007-01-23 (Actual); Study Completion 2007-01-23 (Actual)

PRIMARY OUTCOMES:
Complete virologic response at Month 24 which is normalisation of alanine aminotransferase (ALT) and disappearance of HBV DNA by NAXCOR(brand name of a virus assay kit)

SECONDARY OUTCOMES:
Partial response, histological improvement (at 24 months). Sustained complete response, sustained partial response at 30 months.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, Tehran, Iran